CLINICAL TRIAL: NCT03082768
Title: An Open Label, Brain Positron Emission Tomography, Phase 0 Study of [18F]MNI-968 as a Marker for D1 Receptor in Healthy Subjects
Brief Title: Phase 0 Study of [18F]MNI-968 as a Marker for D1 Receptor in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-968
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
Keywords: HV

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]MNI-968 (Experimental): To evaluate [18F]MNI-968 (aka PF-06730110) as a D1 receptor targeted radiopharmaceutical
  Interventions: Drug: [18F]MNI-968

INTERVENTIONS:
Drug: [18F]MNI-968 — Healthy volunteers recruited for the study will undergo two [18F]MNI-968 injections and PET scans.
  Other Names: PF-06730110

SUMMARY:
The overall goal of this protocol is to evaluate [18F]MNI-968 (aka PF-06730110) as a D1 receptor targeted radiopharmaceutical.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate [18F]MNI-968 (aka PF-06730110) as a D1 receptor targeted radiopharmaceutical.

* To measure the dynamic uptake and washout of [18F]MNI-968 in brain using positron emission tomography (PET) in healthy volunteers.
* To measure blood metabolites of [18F]MNI-968 in the healthy volunteers and to perform invasive as well as non-invasive modeling to assess [18F]MNI-968 binding to D1 receptor.
* To acquire safety data following injection of [18F]MNI-968
* Evaluation of [18F]MNI-968 PET reliability (test/retest) of several outcome measures

ELIGIBILITY:
Inclusion Criteria:

* Are males or females > 18 years of age and < 50 years of age;
* Are in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Are able to communicate well with the investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, they must commit to use a barrier contraception method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for the male subjects for the study duration.
* Male subjects must not donate sperm for the study duration.
* Provide informed consent for study procedures.

Exclusion Criteria:

* Use of any prescription drugs, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing. If needed (i.e. an incidental and limited need), acetaminophen is acceptable, but must be documented as a concomitant medication / significant non-drug therapy.
* Subject has received an investigational therapeutic drug or device within 30 days of screening
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines
* Have a history of blood donation in excess of 500 mL of blood within 30 days prior to screening.
* Have a history or presence of any significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorders which, in the opinion of the investigator, are capable of altering the absorption, metabolism, or elimination of drugs or posing a health risk to participate in the study.
* Have clinically significant findings on laboratory evaluations.
* Have clinically significant findings on ECG evaluation based on cardiology review.
* History of immunodeficiency disease, including a positive HIV test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result.
* History of drug or alcohol abuse within the 12 months prior to screening, or evidence of such abuse as indicated by the laboratory assays conducted during the screening.
* History of tobacco product use within 3 months prior to screening, to be verified by urine cotinine screening.
* Positive pregnancy test result using serum beta-HCG, if female.
* Women who are lactating and breastfeeding.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Tracer uptake will be evaluated in regions of interest for analysis of regional [18F]MNI-968 binding/uptake and expressed in SUV by using established methods for normalization for 7 HV subjects. | 1 year
  Dynamic uptake and washout of [18F]MNI-968 in brain using positron emission tomography (PET) in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Madonia, PA-C, Principal Investigator — Molecular NeuroImaging, LLC
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://mnimaging.com/